CLINICAL TRIAL: NCT05947383
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of up to Two Doses of Psilocybin for the Treatment of Major Depressive Disorder in Adults With Cancer
Brief Title: Two Doses of Psilocybin for the Treatment of MDD in Adults With Cancer
Acronym: 2Dose
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunstone Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUN003
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Major Depressive Disorder
Keywords: psilocybin; cancer; depression
MeSH Terms: conditions — Neoplasms; Depressive Disorder, Major; Depression | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental)
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — Psilocybin 25 mg oral capsule
  Arms: Psilocybin
Drug: Placebo — Niacin 100 mg oral capsule
  Arms: Placebo

SUMMARY:
This is a Phase 2, single-center study to explore the efficacy, safety, and tolerability of up to two 25-mg doses of psilocybin administered at an interval of 9 to 10 weeks in patients with MDD and cancer. This two-part study will administer a fixed dose (25 mg) of psilocybin in a double-blind, randomized, placebo-controlled portion (Dosing Session 1) and subsequently allow rollover into an open-label portion (Dosing Session 2; fixed dose of psilocybin, 25 mg) for patients who do not achieve remission of MDD symptoms after the first dose.

In Dosing Session 1, groups of two to four patients will be randomized, as a cohort, to receive either psilocybin 25 mg or niacin 100 mg (active placebo) in a group session, with each patient supported by their dedicated study therapist and monitored by a second therapist via video feed.

In Dosing Session 2, all eligible participants (i.e., patients who have not achieved remission defined as MADRS < 10 at V7) will receive psilocybin 25 mg in an open-label fashion using the group session model. The study population will include adult men and women who are 18 years of age or older and have diagnoses of both MDD and a malignant neoplasm. MDD is defined as the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) diagnostic criteria for a single or recurrent episode of MDD without psychotic features. A diagnosis of a malignant neoplasm is defined as having a diagnostic code from C00 to C97 according to the International Classification of Diseases, 10th edition (ICD-10). Participants will be recruited through referrals from specialized psychiatric and oncology services as well as through patient self-referrals.

The majority of participants will have no prior exposure to psilocybin or so-called "magic mushrooms"; however, participants with prior recreational experience with psilocybin or "magic mushrooms" are eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF)
2. 18 years of age or above at Screening (V1)
3. Currently meet criteria for MDD (single or recurrent episode as defined by the DSM-5; if single episode, duration of ≥ 3 months) based on medical records, clinical assessment, and documented completion of the Mini International Neuropsychiatric Interview, version 7.0.2 (MINI 7.0.2)
4. A diagnosis of a malignant neoplasm with a diagnostic code from C00 to C97 according to the ICD-10
5. MADRS score ≥ 20 at Screening (V1)
6. Is not currently taking any antidepressant and/or antipsychotic medications or medical cannabis at Screening (V1)
7. Able to complete all protocol-required assessment tools without any assistance or alteration to the copyrighted assessments, and to comply with all study visits
8. Has capacity to consent per judgement of the Investigator

Exclusion Criteria:

1. Current or past history of schizophrenia, psychotic disorder, bipolar disorder, delusional disorder, paranoid personality disorder, schizoaffective disorder, or borderline personality disorder, as assessed by medical history and a structured clinical interview (MINI version 7.0.2)
2. Current (within the past year) alcohol or drug use disorder as defined by the DSM-5 (MINI 7.0.2) at Screening (V1)
3. Significant suicide risk defined by (1) suicidal ideation as endorsed on items 4 or 5 on the C-SSRS within the past year, at Screening, or at Baseline, or; (2) suicidal behaviors within the past year, or; (3) clinical assessment of significant suicidal risk during participant interview
4. Other personal circumstances or behavior judged to be incompatible with establishment of rapport or safe exposure to psilocybin
5. Women who are pregnant, nursing, or planning a pregnancy. Women and men of child-bearing potential and who are sexually active must agree to use an acceptable contraceptive method throughout their participation in the study. Women of child-bearing potential must have a negative urine pregnancy test at Screening (V1) and Baseline (V2)
6. Cardiovascular conditions: recent stroke (< 1 year from signing of ICF), recent myocardial infarction (< 1 year from signing of ICF), uncontrolled hypertension (blood pressure > 140/90), or clinically significant arrhythmia within 1 year of signing the ICF
7. A marked prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 450 ms at screening
8. A history of additional risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome)
9. The use of concomitant medications that prolong the QT/QTc interval
10. Uncontrolled or insulin-dependent diabetes
11. Seizure disorder
12. Positive urine drug screen for illicit drugs or drugs of abuse at V1 and V2. Any positive urine drug test will be reviewed with participants to determine the pattern of use and eligibility will be determined at the Investigator's discretion in conjunction with the medical monitor
13. Current enrollment in any investigational drug or device study or participation in such within 30 days of Screening (V1)
14. Abnormal and clinically significant results on the physical examination, vital signs, ECG, or laboratory tests at Screening (V1) that in the Investigator's opinion may constitute a risk for an individual who is exposed to psilocybin. This includes a value of < 50,000 platelets per cubic millimeter of blood, liver function tests three times the upper limit of normal, and creatine two times above the normal range. Clinically significant abnormal electrolytes or low hemoglobin (< 8 g/L) should be corrected and rechecked prior to enrollment
15. Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, or any other major concurrent illness that, in the opinion of the Investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study
16. Use of psychedelics, including psilocybin but excluding medical marijuana, within the past 6 months and use of psychedelics or cannabis during the current episode of depression
17. Concurrent or recent chemotherapy or radiation therapy that impairs general level of physical functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The Montgomery-Asberg Depression Rating Scale (MADRS) | 8 weeks
  The primary endpoint of efficacy (psilocybin versus active placebo) in this study will be evaluated as change from baseline in MADRS total score at V7 (Week 8).

SECONDARY OUTCOMES:
Treatment-emergent and serious adverse events (TEAEs and SAEs) | 8 weeks
  Incidence and occurrence of treatment-emergent adverse events (TEAEs) and SAEs from the days of psilocybin treatment (V3 and V9) to V7 and V13 and from the day after each psilocybin treatment (V4 and V10) to V7 and V13.
Electrocardiogram (ECG) | 8 weeks
  Incidence of clinically important changes in electrocardiogram (ECG) parameters from Screening (V1) to V7 and from the day before the second psilocybin treatment (V8) to V13.
Laboratory results | 8 weeks
  Incidence of clinically important changes in laboratory results from Screening (V1) to V7 and from V8 to V13.
Vital Signs | 8 weeks
  Incidence of clinically significant changes in vital signs from Screening (V1) to V7 and from V8 to V13.
Columbia Suicide Severity Rating Scale (C-SSRS) | 8 weeks
  Incidence of changes in suicidal ideation/behavior (measured using the Columbia Suicide Severity Rating Scale [C-SSRS]) score at all visits from Baseline (the day before each Dosing Session) (V2 and V8) to V7 and V13.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunstone Medical, PC, Rockville, Maryland, United States